CLINICAL TRIAL: NCT01067898
Title: A Randomized, Double-blind, Placebo-controlled Study on Oral Vitamin D Megadoses - 100 000 or 200 000 IU Vitamin D3 Every Three Months
Brief Title: A Study on Oral Vitamin D Megadoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville-Valtteri Välimäki, MD,PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS-S-D-II; 2009-018139-98 (EudraCT Number); KLnro 1/2010 (Other: The Finnish Medicines Agency Fimea)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Hypovitaminosis D
Keywords: vitamin D supplementation; cholecalciferol; PTH; bone turnover markers; elderly women
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Olive Oil; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 200 000 IU vitamin D3 every three months (Experimental)
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol); Dietary Supplement: calcium carbonate
- 100 000 IU vitamin D3 every three months (Experimental)
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol); Other: olive oil; Dietary Supplement: calcium carbonate
- placebo every three months (Placebo Comparator)
  Interventions: Other: olive oil; Dietary Supplement: calcium carbonate

INTERVENTIONS:
Dietary Supplement: vitamin D3 (cholecalciferol) — vitamin D3 (cholecalciferol) oil 20 000 IU/ml, oral dose of 200 000 IU or 100 000 IU (10ml or 5ml) every three months for one year.
  Other Names: Vigantol vitamin D3 (cholecalciferol) oil 20 000 IU/ml
  Arms: 100 000 IU vitamin D3 every three months; 200 000 IU vitamin D3 every three months
Other: olive oil — 10 ml (placebo group) or 5 ml (100 000 IU vitamin D3 group) oil per os every three months for one year
  Arms: 100 000 IU vitamin D3 every three months; placebo every three months
Dietary Supplement: calcium carbonate — 1000 mg calcium per os every day for one year

SUMMARY:
The purpose of this study is to determine if infrequent administration of oral vitamin D megadoses is effective treatment to maintain serum 25-hydroxyvitamin D(3) above target levels of 50-75 nmol/L. The investigators hypothesize that 100 000 IU or at least 200 000 IU vitamin D3 in every three months would be effective and safe treatment to achieve the target levels.

ELIGIBILITY:
Inclusion Criteria:

* female
* 70-80 yrs old

Exclusion Criteria:

* disease or medication affecting calcium homeostasis
* renal failure (Pt-GFRe-CG < 35 ml/min)

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D3 concentration in relation to the target levels of 50-75 nmol/L | 12 months (including 9 time points)

SECONDARY OUTCOMES:
Decline of creatine clearance (Pt-GFRe-CG) >20% from baseline | 12 months (including 9 timepoints)
Hypercalciuria (dU-Ca >10 mmol/24h) | 12 months (including 9 timepoints)
Hypercalcemia (S-Ca-ion >1,3 mmol/l) | 12 months (including 9 timepoints)
Serum PTH | 12 months (including 9 timepoints)
Serum PINP | 12 months (including 5 timepoints)
Serum CTX | 12 months (including 5 timepoints)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, Department of Medicine, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Pekkarinen T, Valimaki VV, Aarum S, Turpeinen U, Hamalainen E, Loyttyniemi E, Valimaki MJ. The same annual dose of 292000 IU of vitamin D (cholecalciferol) on either daily or four monthly basis for elderly women: 1-year comparative study of the effects on serum 25(OH)D concentrations and renal function. Clin Endocrinol (Oxf). 2010 Apr;72(4):455-61. doi: 10.1111/j.1365-2265.2009.03637.x. Epub 2009 May 25. PMID 19486025
- [Background] Valimaki VV, Loyttyniemi E, Valimaki MJ. Vitamin D fortification of milk products does not resolve hypovitaminosis D in young Finnish men. Eur J Clin Nutr. 2007 Apr;61(4):493-7. doi: 10.1038/sj.ejcn.1602550. Epub 2006 Nov 29. PMID 17136043
- [Background] Valimaki VV, Alfthan H, Lehmuskallio E, Loyttyniemi E, Sahi T, Stenman UH, Suominen H, Valimaki MJ. Vitamin D status as a determinant of peak bone mass in young Finnish men. J Clin Endocrinol Metab. 2004 Jan;89(1):76-80. doi: 10.1210/jc.2003-030817. PMID 14715830